CLINICAL TRIAL: NCT03749499
Title: Targeting of UnControlled Hypertension in Emergency Department (TOUCHED)
Brief Title: Targeting of UnControlled Hypertension in Emergency Department
Acronym: TOUCHED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Heather Prendergast, Professor (CT), Associate Head for Academic Affairs, Resident Research Director, Emergency Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2017-0118; 1R61HL139454-01A1 (NIH)
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Cardiovascular Diseases; Vascular Diseases
Keywords: Emergency Department; Minorities
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases; Emergencies | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research Assistants are blinded to study arm assignment of participant when assessing outcomes measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants randomized to usual care will receive preprinted discharge instructions on HTN and a 48-72-hour referral to our FQHC (or other community health center if pre-assigned though Illinois Medicaid) to schedule their follow-up appointment (current standard of care)
- Educational and Empowerment Intervention (Active Comparator): Participants receive:
  1. HTN Educational Video about high BP, how it is diagnosed, and importance of treatment to prevent secondary complications.
  2. Visual Echocardiogram Image Clips of age/gender-matched echocardiograms will be used to educate and motivate patients to change behavior and improve their BP.
  3. Mobile Health and Remote BP monitoring- participants receive an FDA-approved home blood pressure monitoring (HBPM) kit that includes the Nokia wireless BPM+ monitor and Health Mate mobile app. The app automatically launches when the patient slips on the cuff. Synced data are automatically uploaded from the mobile app to the iCardia server of our study.
  4. A Post-Acute Care HTN Transition consultation (PACHT-c) with a clinical pharmacist or advanced practice nurse (APN).
  Interventions: Other: HTN Educational Video; Other: Visual Echocardiogram Image Clips; Other: Mobile Health and Remote BP monitoring; Other: Post-Acute Care HTN Transition consultation (PACHT-c)

INTERVENTIONS:
Other: HTN Educational Video — The video will educate participants in arm 2 about high BP, how it is diagnosed, and the importance of treating it to prevent secondary complications.
  Arms: Educational and Empowerment Intervention
Other: Visual Echocardiogram Image Clips — Visual clips of age/gender-matched echocardiograms will be used to educate and motivate patients to change their behavior and improve their BP. We have found that real time visualization of cardiac ultrasound images with active discussion of findings is a significant patient motivator and empowerment tool, and was a significant factor in the success of our previous pilot study.
  Arms: Educational and Empowerment Intervention
Other: Mobile Health and Remote BP monitoring — All participants randomized to the intervention group will receive an FDA-approved HBPM kit that includes the Nokia wireless (self-inflating) BPM+ monitor and Health Mate mobile app. The app automatically launches when the patient slips on the cuff and turns on the monitor to measure his/her BP. Synced data are automatically uploaded from the mobile app to the iCardia server of our study.
  Arms: Educational and Empowerment Intervention
Other: Post-Acute Care HTN Transition consultation (PACHT-c) — All participants randomized to the E2 intervention will have a focused consultation with either a clinical pharmacist or an APN. During this consultation, the pharmacist/APN repeats the BP measurement; reviews the screening assessments; and reviews general principles of BP control including nutrition, exercise, and smoking cessation. BP will be managed according to the current published guidelines available at the time of funding regarding initiation of first-line antihypertensive medications. Patients with BP ≥160/100 mmHg may be started on antihypertensive medications by the provider during the consultation if appropriate.
  Arms: Educational and Empowerment Intervention

SUMMARY:
The proposed project underscores the following: 1) The prevalence of uncontrolled/undiagnosed hypertension (HTN) in underrepresented groups presenting to the ED is alarmingly high, and 2) ED engagement and early risk assessment/stratification is a cost-effective, feasible innovation to help close health disparity gaps in HTN. This proposal involves a two-arm randomized controlled trial of up to 770 patients from the Emergency Department at University of Illinois Hospital with elevated blood pressure (BP). The primary objective is to determine the effectiveness of an emergency department-initiated Educational and Empowerment (E2) intervention with a Post Acute Care Hypertension Consultation (PACHT-c) intervention (arm 2) on the primary outcome of mean systolic blood pressure (SBP) differences between the two trial arms at 6-months post intervention. Secondary objectives include evaluating the effectiveness of this ED education and empowerment intervention on mean SBP and diastolic blood pressure (DBP) differences at 3-months, and mean DBP differences at 6-months.

DETAILED DESCRIPTION:
The study is a single-site randomized controlled trial (RCT) focused on a high-risk ED population with evidence of moderately elevated BP (≥140/90 mmHg) at discharge. ED patients will be recruited and randomized into two arms: 1) usual care (preprinted discharge instructions and 48-72 hour referral to a federally qualified health center (FQHC) or assigned provider as appropriate); 2) ED-initiated E2 intervention program followed by 48-72 hour referral to a FQHC (or assigned health center). Based on the ED population demographics (70% ethnic minorities), the majority of participants will be underrepresented minorities (NHB and Hispanic) and low-income individuals. The investigators propose the following specific aims and hypotheses:

Aim 1: Evaluate the effectiveness of an ED-based E2 + PACHT-c intervention (arm 2) on the primary outcome of mean SBP difference at 6-months post-intervention compared to usual care (arm 1).

H1: The mean SBP difference (from baseline) will be significantly greater in the E2+ PACHT-c group (arm 2) compared to the usual care group (arm 1) at 6- months post-randomization, i.e., SBP change in arm 2 > arm 1 at 6-months post-randomization.

Aim 2: Evaluate the effectiveness of an ED-based E2 intervention with PACHT-c on the secondary outcome of mean SBP and DBP differences at 3-months, and mean DBP differences at 6 months post-intervention compared to usual care.

H2: The mean SBP and DBP differences from baseline to 3- months post-intervention and mean DBP at 6-months post intervention will be significantly greater in the ED-based E2 intervention compared to the usual care group, i.e., SBP and DBP change in arm 2 > arm 1 at 3 -months post-intervention and DBP change in arm 2 > arm 1 at 6 -months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* BP>=140/90 and <=180/110 mm Hg at time of discharge from ED
* Verbal fluency in English or Spanish
* Age 18-75 years

Exclusion Criteria:

* Unable to verbalize comprehension of study, impaired decision-making or documented dementia
* Plans to move from Chicago area within the next year
* Pregnant or trying to get pregnant
* COVID-19 positive within the past 14 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Prendergast, MD, MPH, MS, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The TOUCHED data sets will be submitted to the NHLBI Data repository, and will include the following:
  * Data Information collected and recorded from study participants, including baseline, interim visit, ancillary data, outcome data, laboratory measurements not otherwise summarized, blood pressure measurements; quantitative results from survey assessments; clinical event surveillance and follow-up contacts.
  * Study documentation: Descriptive information regarding the conduct of the study and collection of Data, including study protocol, manual of operations/procedures, annotated data collection forms, codebooks /data dictionary, and descriptions of data derived from procedures.
  In the preparation and delivery of the Data to the NHLBI Data Repository, all personal identifiers will be eliminated. A summary of all proposed modifications and deletions to be made to a data set will be submitted to and approved by the NHLBI Data Repository representative prior to their implementation.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The TOUCHED data set will be submitted to the NHLBI Program Officer, no later than 3 years after the end of the clinical activity (final patient follow-up, etc.) or 2 years after the main paper of the trial has been published, whichever comes first.

REFERENCES:
- [Derived] Prendergast H, Kitsiou S, Petzel Gimbar R, Freels S, Sanders A, Daviglus M, Kotini-Shah P, Carter B, Del Rios M, Heinert S, Khosla S. Emergency Department-Based Education and mHealth Empowerment Intervention for Hypertension: The TOUCHED Randomized Clinical Trial. JAMA Cardiol. 2025 Jul 1;10(7):657-665. doi: 10.1001/jamacardio.2025.0675. PMID 40266598
- [Derived] Prendergast HM, Petzel-Gimbar R, Kitsiou S, Del Rios M, Lara B, Jackson M, Heinert S, Carter BL, Durazo-Arvizu RA, Daviglus M. Targeting of uncontrolled hypertension in the emergency department (TOUCHED): Design of a randomized controlled trial. Contemp Clin Trials. 2021 Mar;102:106283. doi: 10.1016/j.cct.2021.106283. Epub 2021 Jan 20. PMID 33484897

RESULTS

PARTICIPANT FLOW:
Groups:
- Educational and Empowerment Intervention: Participants receive:
  1. HTN Educational Video about high BP, how it is diagnosed, and importance of treatment to prevent secondary complications.
  2. Visual Echocardiogram Image Clips of age/gender-matched echocardiograms will be used to educate and motivate patients to change behavior and improve their BP.
  3. Mobile Health and Remote BP monitoring- participants receive an FDA-approved home blood pressure monitoring (HBPM) kit that includes the monitor and Health Mate mobile app. The app automatically launches when the patient slips on the cuff. Synced data are automatically uploaded from the mobile app to the iCardia server of our study.
  4. A Post-Acute Care HTN Transition consultation (PACHT-c) with a clinical pharmacist or advanced practice nurse (APN).
  Post-Acute Care HTN Transition consultation (PACHT-c): All participants randomized to the E2 intervention will have a focused consultation with either a clinical pharmacist or an APN. During this consultation, the pharmacist/APN repeats the BP measurement; reviews the screening assessments; and reviews general principles of BP control including nutrition, exercise, and smoking cessation. BP will be managed according to the current published guidelines available at the time of funding regarding initiation of first-line antihypertensive medications. Patients with BP ≥160/100 mmHg may be started on antihypertensive medications by the provider during the consultation if appropriate.
Period: Overall Study
Arm/Group | Usual Care | Educational and Empowerment Intervention
Started | 285 | 289
Completed | 203 | 210
Not Completed | 82 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Educational and Empowerment Intervention | Total
Number analyzed (Participants) | 285 | 289 | 574
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (13) | 50.3 (11.9) | 51.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 161 | 323
  Male | 123 | 128 | 251
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 10 | 27
  Black | 204 | 209 | 413
  Hispanic/Latino | 56 | 59 | 115
  Other | 8 | 11 | 19
Insurance [Count of Participants; unit: Participants]
  Private | 69 | 85 | 154
  Medicare/Medicaid | 149 | 135 | 284
  Other | 7 | 8 | 15
  Unknown/Missing | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Mean Systolic Blood Pressure (SBP) Difference at 6 Months Post-intervention Compared to Usual Care.
Description: Blood pressure will be collected at two time points (baseline and 6 months). ED-pharmacists and trained research assistants will perform BP measurements using standardized procedures.
Time Frame: Baseline, 6 months after baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care | Educational and Empowerment Intervention
Number analyzed (Participants) | 203 | 210
mmHg | -9.2 (24.4) | -14.0 (19.3)

2. Secondary Outcome: Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Differences at 3 Months Post-intervention Compared to Usual Care.
Description: Blood pressure will be collected at two time points (baseline and 3 months). ED-pharmacists and trained research assistants will perform BP measurements using standardized procedures.
Time Frame: Baseline, 3 months after baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care | Educational and Empowerment Intervention
Number analyzed (Participants) | 151 | 157
mmHg
  SBP | -9.8 (22.5) | -14 (20.5)
  DBP | -1.5 (13.4) | -2.4 (11.7)

3. Secondary Outcome: Diastolic Blood Pressure (DBP) Difference at 6 Months Post-intervention Compared to Usual Care.
Description: as for outcome 1
Time Frame: Baseline, 6 months after baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care | Educational and Empowerment Intervention
Number analyzed (Participants) | 203 | 210
mmHg | -1.3 (14.5) | -3.3 (12.1)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Groups:
- Educational and Empowerment Intervention: Participants receive:
  HTN Educational Video about high BP, how it is diagnosed, and importance of treatment to prevent secondary complications.
  Visual Echocardiogram Image Clips of age/gender-matched echocardiograms will be used to educate and motivate patients to change behavior and improve their BP.
  Mobile Health and Remote BP monitoring- participants receive an FDA-approved home blood pressure monitoring (HBPM) kit that includes the monitor and Health Mate mobile app. The app automatically launches when the patient slips on the cuff. Synced data are automatically uploaded from the mobile app to the iCardia server of our study.
  A Post-Acute Care HTN Transition consultation (PACHT-c) with a clinical pharmacist or advanced practice nurse (APN).
  Post-Acute Care HTN Transition consultation (PACHT-c): All participants randomized to the E2 intervention will have a focused consultation with either a clinical pharmacist or an APN. During this consultation, the pharmacist/APN repeats the BP measurement; reviews the screening assessments; and reviews general principles of BP control including nutrition, exercise, and smoking cessation. BP will be managed according to the current published guidelines available at the time of funding regarding initiation of first-line antihypertensive medications. Patients with BP ≥160/100 mmHg may be started on antihypertensive medications by the provider during the consultation if appropriate.
Arm/Group | Usual Care | Educational and Empowerment Intervention
All-Cause Mortality (participants affected / at risk) | 7/285 | 0/289
Serious Adverse Events (participants affected / at risk) | 0/285 | 0/289
Other Adverse Events (participants affected / at risk) | 0/285 | 0/289

LIMITATIONS AND CAVEATS:
Recruitment and retention during the pandemic posed challenges to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03749499/Prot_SAP_000.pdf